CLINICAL TRIAL: NCT01440868
Title: SLI STUDY: Sustained Lung Inflation in the Delivery Room in Preterm Infants at High Risk of Respiratory Distress Syndrome. A RCT Study
Brief Title: Sustained Lung Inflation in the Delivery Room in Preterm Infants at High Risk of Respiratory Distress Syndrome
Acronym: SLIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Carlo Dani, Associate Professor of Pediatrics, University of Florence
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-2011
Record Dates: First submitted 2011-09-16; First posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome, Newborn; Delivery Rooms; Resuscitation; Premature Birth; Infant, Newborn; Respiration, Artificial
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Distress Syndrome, Newborn; Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SLI group (Experimental): In this group the preterm infants will receive sustained lung inflation (SLI) with mask in the delivery room
  Interventions: Procedure: Sustained lung inflation
- Control (No Intervention): Preterm infants will be assisted in the delivery room without sustained lung inflation.

INTERVENTIONS:
Procedure: Sustained lung inflation — Sustained lung inflation (SLI) will be performed with mask using a pressure control system (Neopuff, Fisher & Paykel, Inc). Peak inflation pressure (PIP) of 25 cm H2O will be delivered for 15 seconds and then reduced to a PEEP of 5 cm H2O. A second SLI manoeuvre will be repeated in case of persistent hearth failure (HR <100 bpm ).
  Other Names: Lung recruitment
  Arms: SLI group

SUMMARY:
BACKGROUND. Sustained lung inflation (SLI) associated to an adequate PEEP may help the efficacy of the respiratory effort in lung of preterm infants at risk for respiratory distress syndrome (RDS) and reduce need of mechanical ventilation (MV).

The investigators aim will be to demonstrate the hypothesis that the introduction of SLI in the delivery room protocol may reduce the need of MV in preterm infants.

STUDY DESIGN: Multicenter prospective randomized controlled trial. The study will be carried out at the neonatal care units of the Careggi Infants with a gestational age between 25 and 28 weeks will be eligible and randomized at birth to receive SLI or not. Peak inflation pressure (PIP) of 25 cm H2O will be delivered for 15 seconds and then reduced to a positive end expiratory pressure (PEEP) of 5 cm H2O.

Primary endpoint will be the need of MV within the first 72 hrs of life (excluding the transient tracheal intubation for surfactant replacement: e.g. INSURE). Population size: hypothesizing that SLI maneuver might decrease the need of MV during the first 72 hours of life from 35 to 20% the investigators calculated that 138 newborns must be enrolled in each groups to detect this difference statistically significant with 80% power at 0.05 level.

DETAILED DESCRIPTION:
BACKGROUND Sustained lung inflation (SLI) applied at birth in the delivery room has been demonstrated to lead to clearance of lung fluid and achievement of a precocious functional residual capacity (FRC) both in animal and human studies. SLI associated to an adequate positive end expiratory pressure (PEEP) may help the efficacy of the respiratory effort in lung of preterm infants at risk for respiratory distress syndrome (RDS) and reduce need of mechanical ventilation (MV).

OBJECTIVES Our aim will be to demonstrate the hypothesis that the introduction of SLI in the delivery room protocol may reduce the need of MV in the first 72 hours of life in preterm infants at risk for RDS improving their respiratory outcome.

STUDY DESIGN This is a multicenter prospective randomized controlled trial. The study will be carried out at the neonatal care units of the Careggi University Hospital of Florence, the "V. Buzzi" Children Hospital of Milan, IRCCS Ospedale Maggiore Policlinico of Milan,the Catholic University of the Sacred Heart of Rome, the "S. Giovanni" Hospital of Rome, the Regional Hospital of Bozen, the Hospital of Varese, the the Sant'Anna University Hospital of Pisa, the "Maggiore" Hospital of Bologna, the "Di Venere" Hospital of Bari, the University Hospital of Foggia.

Inborn infants with a gestational age between 25 and 28 weeks will be eligible and randomized at birth in two groups. Group A: (SLI group) in this group the preterm infants will receive SLI with mask for initial alveolar recruitment using a pressure control system (Neopuff, Fisher & Paykel, Inc) in addition to American Academy of Pediatrics (AAP) guidelines for neonatal resuscitation. Peak inflation pressure (PIP) of 25 cm H2O will be delivered for 15 seconds and then reduced to a PEEP of 5 cm H2O. A second SLI manoeuvre will be repeated in case of persistent hearth failure (HR <100 bpm.Group B (control group: in this group the preterm infants will be resuscitated at birth according to AAP guidelines without SLI manoeuvre.

Infants in both the groups who will not be able to reach a good respiratory and/or cardiac effort, they will undergo tracheal intubation to start MV. Then, in neonatal intensive care unit (NICU), infants who will continue to breath spontaneously will be supported by nasal continuous positive airway pressure (NCPAP), bi-level positive airway pressure (BiPAP) or nasal intermittent mandatory ventilation (N-IMV) (PEEP at 5-7 cmH2O). Surfactant (Curosurf ®, Chiesi, Parma, Italia) will be administered (200 mg/kg) to newborns with FiO2 >0.40 or mechanically ventilated. MV will be started if blood pH <7.20, PCO2 >65 mm Hg, pO2 <50 mm Hg with a fraction of inspired oxygen (FiO2) >0.50 or in case of severe apnea; the objective of MV will be to maintain a PaCO2 45-65 mmHg and a PaO2 50-75 mmHg. Preterm infants will be extubated from MV when airway pressure will be <7 cmH2O, FiO2 <0.30, and in absence of severe apnea after caffeine therapy. After extubation it will be allowed to support infant with oxygen-therapy, NCPAP, BiPAP or N-IMV.

ENDPOINTS. Primary endpoint will be the need of MV within the first 72 hrs of life [(excluding the transient tracheal intubation for surfactant replacement: e.g. Intubation-SURfactant-Extubation (INSURE)]. Success criteria will be the lack of MV in the first 72 hrs of life. Secondary endpoints will be the occurrence of MV >3 hrs of life, length of MV and other non invasive respiratory supports (NCPAP/BiPAP/N-IMV), need of surfactant and number of doses, mortality, occurrence of bronchopulmonary dysplasia (BPD:oxygen-therapy at 36 post- conceptional age), intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), retinopahty of prematurity (ROP) and necrotizing enterocolitis (NEC), sepsis, and length of NICU and hospital stay.

STATISTICAL ANALYSIS. Failure of treatment will be considered the need of MV during the first 72 hrs of life in both groups.

Population size: hypothesizing that SLI maneuver might decrease the need of MV during the first 72 hours of life from 35 to 20% we calculated that 138 newborns must be enrolled in each groups to detect this difference statistically significant with 80% power at 0.05 level.

Clinical characteristics of the two groups will be described by mean values and standard deviation, or median values and range, or by rate and percentage. The t-test, Wilcoxon rank-sum test, and Fisher's exact test will be used to compare continuous normally distributed data, nonparametric continuous data, and categorical data, respectively.

Multiple regression analysis will be performed to assess the possible influence of confounding variables (i.e.: gestational age, birth weight, etc.) on the primary endpoint predictive factors. Effect estimates will be expressed as relative risk (RR) with profile likelihood-based 95% confidence limits.

ELIGIBILITY:
Inclusion Criteria:

* parental informed consent
* gestational age 25-28 weeks

Exclusion Criteria:

* fetal hydrops
* major congenital malformation
* inherited metabolic diseases

Max Age: 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Need of mechanical ventilation | First 72 hrs of life
  Preterm infants are at risk of developing respiratory distress syndrome requiring mechanical ventilation. Sustained lung inflation in the delivery room might contribute to decrease the need of mechanical ventilation during the first 72 hrs of life because later other factors (i.e.: sepsis)than prematurity itself could induce this need.

SECONDARY OUTCOMES:
Complication rate | Participants will be followed for the duration of hospital stay, an expected average of 13 weeks
  We will evaluate the occurrence of mechanical ventilation (MV) >3 hrs of life, length of MV and other non invasive respiratory supports, need of surfactant, mortality, the occurrence of the main prematurity complication such as bronchopulmonary dysplasia (BPD), intraventricular hemorrhage (IVH) , periventricular leukomalacia (PVL), retinopathy of prematurity (ROP) and necrotizing enterocolitis (NEC), sepsis, and length of neonata intensive care (NICU) and hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Dani, MD, Study Chair — University of Florence, Italy
Locations (1):
- Department of Surgical and Medical Critical Care, Unversity of Florence, Florence, Italy

REFERENCES:
- [Derived] Dani C, Lista G, Pratesi S, Boni L, Agosti M, Biban P, Del Vecchio A, Gazzolo D, Gizzi C, Magaldi R, Messner H, Mosca F, Sandri F, Scopesi F, Trevisanuto D, Vento G. Sustained lung inflation in the delivery room in preterm infants at high risk of respiratory distress syndrome (SLI STUDY): study protocol for a randomized controlled trial. Trials. 2013 Mar 8;14:67. doi: 10.1186/1745-6215-14-67. PMID 23497495